CLINICAL TRIAL: NCT02624310
Title: A Phase II, Randomized, Double Blind, Cross-over, Placebo-controlled Study on Norepinephrine Replenishment Therapy Using L-DOPS in Congenital Insensitivity to Pain With Anhidrosis Patients
Brief Title: A Study of Norepinephrine in Patients With Congenital Insensitivity to Pain and Anhidrosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14-01774
Record Dates: First submitted 2014-09-30; First posted 2015-12-08 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: HSAN Type IV
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Droxidopa First, Placebo Second (Experimental): Participants in this arm will receive droxidopa first, then cross over and receive placebo
  Interventions: Drug: Droxidopa (L-DOPS); Drug: Placebo
- Placebo First, Droxidopa Second (Experimental): Participants in this arm will receive placebo first, then cross over and receive droxidopa
  Interventions: Drug: Droxidopa (L-DOPS); Drug: Placebo

INTERVENTIONS:
Drug: Droxidopa (L-DOPS) — Patients will be given their initial 100 mg of L-DOPS (visit 2a). The dose of L-DOPS will be increased in escalation in the following visits. Each day the dose will be increased 100 mg. The escalating doses of L-DOPS will be 200 mg (visit 2b), 300 mg (visit 2c), 400 mg (visit 2d), 500 mg (visit 2e) and 600 mg (visit 2f). Following this titration step, L-DOPS will be withdrawn from the subjects for a minimum of two weeks, when the subject will return for visit 3.Visit 3a,b,c,d,e,f: Carbidopa open-label dose titration. This titration step will be similar than L-DOPS titration. Carbidopa starting dose will be 100 mg (visit 3a) and will be increased 100 mg each visit up to a maximum of 600 mg (visit 3f). Following carbidopa titration step, patients will be withdrawn from the drug for minimum of two weeks, then the subject will return for the next titration step (visit 4).
  Other Names: Northera
Drug: Placebo

SUMMARY:
The aim of this study is to increase norepinephrine levels in a population of young adults where NE levels are very low or undetectable. In order to achieve this, the optimal dose will be determined in a titration step. In the titration step, different doses of L-DOPS will be tested in order to find the optimal and safest dose suitable for each individual enrolled in the study. Because L-DOPS has never been used in the US in children or young adults, with this titration step investigators will also determine the safest dose for this population.

Currently, L-DOPS is being used in our center to treat othostatic hypotension in autonomic failure. The titration step for this study starts with the dose of 100 mg and increases in an escalating manner up to a maximum of 600 mg a day (see investigational brochure attached).

L-DOPS has been developed in capsules for oral used and all the previous safety data has been performed using this route. Oral route is the one that will used during study.

Carbidopa is well tolerated, safe in children and it has been used in this population in the US without severe adverse effects.

DETAILED DESCRIPTION:
CIPA patient do have very low or undetectable levels of norepinephrine in plasma and also have significant cognitive and behavioral problems. The aim of this project is to increase NE levels in brain and evaluate if this increase improve cognitive cognition or behavior.

Both drugs from the study have never been used in CIPA patients before, it is therefore very important to evaluate safety and tolerability of L-DOPS and carbidopa in this population.

Even if NE levels are very low in plasma of CIPA subjects, it is not know if NE levels are also low in central nervous system. It is very likely that this is also the case, however, levels of NE in brain will be checked in one CIPA subject as a prof of concept.

Study overview: Patients with CIPA will be screened and enrolled (visit 1) into part 1 of the pilot trial. Safety parameters including, adverse events, blood chemistries for renal and liver function testing, 12 lead electrocardiogram, temperature, weight and blood pressure (supine, seated and standing), non-verbal intelligence and behavior test, 24 hour urinary catecholamine excretion and plasma dopamine levels will be measured at baseline.

The patients will enter an open-label dose titration phase (visit 2a,b,c,d,e,f) during which adverse events will be continuously monitored. After reaching a dose the 100 mg/day dose, patients will be questioned about adverse events and have their blood pressure (supine, sitting and standing) measured. If no adverse events or abnormalities are detected patients will continue the dose titration. Safety assessments will be repeated and safety bloods obtained when the patient reaches the maximum tolerated dose.

After completion of the dose titration, patients who are able to tolerate L-DOPS will enter into a second open-label dose titration phase where carbidopa will be titrated (visit 3a,b,c,d,e,f). A period of two weeks will be allowed to washout the L-DOPS before starting with the carbidopa titration.

Carbidopa have been previously used in clinical studies in children, young adults and adults in our group and no adverse effects have been reported. There is no reason to think that carbidopa may be unsafe in CIPA patients, however, the aim of these titration step is to check safety and tolerability of the drug in this population. Subjects will receive a dose of 100 mg/day and will be questioned about adverse events and have their blood pressure (supine, sitting and standing) measured. If no adverse events or abnormalities are detected patients will continue the dose titration. In the following steps, the doses of carbidopa will be increased 100 mg daily up to a total of 600 mg/day. Safety assessments will be repeated and safety bloods obtained when the patient reaches a total daily dose of 600 mg/day.

In the final phase of the titration, both L-DOPS and carbidopa will be administered (visit 4a,b,c,d,e). The starting dose of L-DOPS will be the maximum tolerated dose during the L-DOPS titration step. The dose of carbidopa that will be administered with L-DOPS will be the maximum tolerated dose. L-DOPS will be increase in 100 mg/day up to 600 mg/day, unless any adverse affect is observed and then the titration will stop at that dose of L-DOPS. The dose of carbidopa will be the maximum tolerated during the titration and will not be increased.

After reaching the maximum L-DOPS/carbidopa tolerated dose, patients will be questioned about adverse events with the medication and have their blood pressure (supine, sitting and standing) measured. After the safety evaluation if no adverse events or abnormalities are observed in the patients will continue with the study. A period of two weeks will be allowed to washout the L-DOPS/carbidopa before starting with placebo-controlled double-blind cross over phase.

Patients who successfully complete titration will proceed to the randomized placebo control phase. Before proceeding to this part, researcher will review of safety data from the titration. Patients will be randomized in a double-blind fashion, to receive either L-DOPS/carbidopa or matching placebo. Patients will take the medication for 4 weeks.

After 4 weeks, 24 urinary catecholamine excretion, plasma dopamine levels, behavior scores, safety parameters and adverse events will be measured (visit 5), before patients are crossed over (visit 6). A similar dose withdrawal scheme will be implemented to prevent adverse effects from acute withdrawal. Patients will be followed for a further 4-weeks. After completion of the cross over period, patients will undergo final evaluation (visit 7) during which safety and efficacy measures will be repeated. To conclude the study, 2 weeks after completing the pilot-trial, patients will receive a follow up phone call to monitor any adverse events.

All necessary safety information will be reported to the FDA in accordance with 312.32 IND safety reports as outlined in Title 21 Food and Drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 15 years old or older
* Patient carrying the genetic mutation for the NTRK1 gene
* Patients (or guardian if patient it is underage) have signed a written consent to participate in the study after being fully informed about the procedure of the study and their right to withdraw at anytime during it.

Exclusion Criteria:

* Patients taking amphetamines, norepinephrine reuptake inhibitors.
* Patients taking any medication that can interact with the study drug L- DOPS.
* Patients with previous severe hypertension (systolic blood pressure >170 mmHg)
* Patients with arrhythmias or any other cardiac condition.
* Women who are pregnant or breast feeding
* Have a renal or hepatic disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 8 weeks
  Safety and tolerability will be assessed using general physical and neurological examinations, vital signs including blood pressure and heart rate, temperature and body weight, blood chemistries including serum creatinine, electrolytes, transaminases and liver function tests, 12 lead electrocardiograms and adverse events monitoring.